CLINICAL TRIAL: NCT03149042
Title: Validation of a Computed Tomography (CT) Based Fractional Flow Reserve (FFR) Software Using the 320 Detector Aquilion ONE CT Scanner.
Status: Completed | Type: Observational
Sponsor: State University of New York at Buffalo (Other)
Responsible Party: Principal Investigator, Ciprian Ionita, Principal Investigator, State University of New York at Buffalo
Other Study IDs: 01
Record Dates: First submitted 2017-05-08; First posted 2017-05-11 (Actual); Results first posted 2020-06-23 (Actual); Last update posted 2020-11-17 (Actual); Status verified 2020-11

CONDITIONS: Atherosclerosis, Coronary
Keywords: FFR; Fractional Flow Reserve; Atherosclerosis; Coronary; stenosis
MeSH Terms: conditions — Coronary Artery Disease; Atherosclerosis; Constriction, Pathologic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- CCTA: Patients who are scheduled for clinically mandated elective invasive coronary angiography (ICA) at Buffalo General Hospital.
  Interventions: Diagnostic Test: CCTA

INTERVENTIONS:
Diagnostic Test: CCTA — Diagnostic Test

SUMMARY:
Coronary Computed Tomography Angiography (CCTA) contrast opacification gradients and FFR-CT estimation can aid in the severity estimation of significant atherosclerotic lesions. Currently, FFR-CT algorithms can only be optimized using theoretical models and can only be validated in large multi-center clinical trials. Using patient specific 3D printed coronary phantoms would allow optimization of FFR-CT algorithms with a measured validation technique without the need for large clinical trials. Thus the investigators believe that this study will result in a FFR-CT algorithm/method with a better predictability for arterial lesion severity than those existing on the market today. Flow measurements will be compared with: CT-FFR for both patients and phantoms, angio lab FFR measurements and 30 days follow-up. This pilot clinical study includes ~50 patients over a year and half at GVI.

DETAILED DESCRIPTION:
Coronary Computed Tomography Angiography (CCTA) contrast opacification gradients and FFR-CT estimation can aid in the severity estimation of significant atherosclerotic lesions. Following this trend, the investigators recently developed a collaboration between Brigham and Women's Hospital (BWH) and Gates Vascular Institute (GVI). The investigators 3D-printed patient specific coronary phantoms at (GVI) and scanned them with a Toshiba Aquilion scanner to test several aspects of the contrast opacification gradients using a method established at BWH. The initial results showed strong correlation between the flow in the phantom and opacification gradients. The investigators believe that this approach could be further developed to test and validate FFR-CT algorithms. Currently, FFR-CT algorithms can only be optimized using theoretical models and can only be validated in large multi-center clinical trials. This phantom approach would allow optimization of FFR-CT algorithms with a measured validation technique without the need for large clinical trials. Thus the investigators believe that this study will result in a FFR-CT algorithm/method with a better predictability for arterial lesion severity than those existing on the market today. The approach is to use the infrastructure at GVI to perform a detailed validation of the FFR-CT method using 3D printed patient specific phantoms. The subject enrollment criteria is: at least one CCTA, at least one lesion with >50% stenosis or 30-50% and an angio based FFR. Each patient will have a 3D phantom printed, containing the culprit lesion and used in a benchtop flow analysis. Flow measurements will be compared with: CT-FFR for both patients and phantoms, angio lab FFR measurements and 30 days follow-up. This pilot clinical study will include ~50 patients over a year and half at GVI. The investigators are confident that this approach performed via 3D-phantom testing will prove the validity of FFR-CT based measurements as well as develop a new standard for validating FFR-CT algorithms.

ELIGIBILITY:
Inclusion Criteria:

* All the patients >18 yrs of age , who are undergoing CCTA and angio-FFR. Patients who are (1) scheduled for clinically mandated elective invasive coronary angiography (ICA) at Buffalo General Hospital or (2) clinically mandated CTA will be screened.

Exclusion Criteria:

* Adults unable to consent
* Individuals who are not yet adults (infants, children, teenagers)
* Pregnant women
* Prisoners
* atrial fibrillation,
* Renal insufficiency (estimated glomerular filtration rate (GFR) <60 ml/min/1.73 m2),
* Active Bronchospasm prohibiting the use of beta blockers
* Morbid obesity (body mass index 40 kg/m2)
* Contraindications to iodinated contrast.
* Emergencies requiring immediate intervention or patients unable to consent.
* Patients not showing coronary calcium during Calcium Scoring procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are (1) scheduled for clinically mandated elective invasive coronary angiography (ICA) at Buffalo General Hospital or Juntendo Hospital Japan (2) clinically mandated CTA will be screened.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2016-05-28 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2019-04-21 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical and Translational Research Center Room 8052, Buffalo, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sommer K, Izzo RL, Shepard L, Podgorsak AR, Rudin S, Siddiqui AH, Wilson MF, Angel E, Said Z, Springer M, Ionita CN. Design Optimization for Accurate Flow Simulations in 3D Printed Vascular Phantoms Derived from Computed Tomography Angiography. Proc SPIE Int Soc Opt Eng. 2017 Feb 11;10138:101380R. doi: 10.1117/12.2253711. Epub 2017 Mar 13. PMID 28663663
- [Background] Ionita, C., Angel, E., Mitsouras, D., Rudin, S., Bednarek, D., Zaid, S., Wilson, M. and Rybicki, F. (2016), TU-H-CAMPUS-IeP2-03: Development of 3D Printed Coronary Phantoms for In-Vitro CT-FFR Validation Using Data from 320- Detector Row Coronary CT Angiography. Med. Phys., 43: 3781. doi:10.1118/1.4957681
- [Background] Kelsey N. Sommer, Lauren M. Shepard, Vijay Iyer, Erin Angel, Michael F. Wilson, Frank J. Rybicki, Dimitrios Mitsouras, Kanako Kunishima Kumamaru, Stephen Rudin, and Ciprian N. Ionita. Comparison of benchtop pressure gradient measurements in 3D printed patient specific cardiac phantoms with CT-FFR and computational fluid dynamic simulations, Proc. SPIE 10953, Medical Imaging 2019: Biomedical Applications in Molecular, Structural, and Functional Imaging, 109531P (15 March 2019);
- [Background] Shepard LM, Sommer KN, Angel E, Iyer V, Wilson MF, Rybicki FJ, Mitsouras D, Molloi S, Ionita CN. Initial evaluation of three-dimensionally printed patient-specific coronary phantoms for CT-FFR software validation. J Med Imaging (Bellingham). 2019 Apr;6(2):021603. doi: 10.1117/1.JMI.6.2.021603. Epub 2019 Mar 12. PMID 30891468
- [Background] Sommer KN, Shepard L, Karkhanis NV, Iyer V, Angel E, Wilson MF, Rybicki FJ, Mitsouras D, Rudin S, Ionita CN. 3D Printed Cardiovascular Patient Specific Phantoms Used for Clinical Validation of a CT-derived FFR Diagnostic Software. Proc SPIE Int Soc Opt Eng. 2018 Feb;10578:105780J. doi: 10.1117/12.2292736. Epub 2018 Mar 12. PMID 29899591
- [Background] Shepard L, Sommer K, Izzo R, Podgorsak A, Wilson M, Said Z, Rybicki FJ, Mitsouras D, Rudin S, Angel E, Ionita CN. Initial Simulated FFR Investigation Using Flow Measurements in Patient-specific 3D Printed Coronary Phantoms. Proc SPIE Int Soc Opt Eng. 2017 Feb 11;10138:101380S. doi: 10.1117/12.2253889. Epub 2017 Mar 13. PMID 28649159
- [Background] Kelsey N. Sommer, Lauren M. Shepard, Vijay Iyer, Erin Angel, Michael F. Wilson, Frank J. Rybicki, Dimitrios Mitsouras, Ciprian Ionita. Study of the effect of boundary conditions on fractional flow reserve using patient specific coronary phantoms. Proceedings Volume 11317, Medical Imaging 2020: Biomedical Applications in Molecular, Structural, and Functional Imaging; 113171J (2020) https://doi.org/10.1117/12.2548472
- [Result] Sommer KN, Shepard LM, Mitsouras D, Iyer V, Angel E, Wilson MF, Rybicki FJ, Kumamaru KK, Sharma UC, Reddy A, Fujimoto S, Ionita CN. Patient-specific 3D-printed coronary models based on coronary computed tomography angiography volumes to investigate flow conditions in coronary artery disease. Biomed Phys Eng Express. 2020 May 14;6(4):045007. doi: 10.1088/2057-1976/ab8f6e. PMID 33444268
- [Result] Kumamaru KK, Angel E, Sommer KN, Iyer V, Wilson MF, Agrawal N, Bhardwaj A, Kattel SB, Kondziela S, Malhotra S, Manion C, Pogorzelski K, Ramanan T, Sawant AC, Suplicki MM, Waheed S, Fujimoto S, Sharma UC, Rybicki FJ, Ionita CN. Inter- and Intraoperator Variability in Measurement of On-Site CT-derived Fractional Flow Reserve Based on Structural and Fluid Analysis: A Comprehensive Analysis. Radiol Cardiothorac Imaging. 2019 Aug 29;1(3):e180012. doi: 10.1148/ryct.2019180012. eCollection 2019 Aug. PMID 33778507
- See also: results — https://iopscience.iop.org/article/10.1088/2057-1976/ab8f6e/meta

RESULTS

PARTICIPANT FLOW:
Groups:
- CCTA: Patients who are scheduled for clinically mandated elective invasive coronary angiography (ICA) at Buffalo General Hospital.
  CCTA (Coronary CT angiography) Diagnostic Test
Period: Overall Study
Arm/Group | CCTA
Started | 75
Completed | 52
Not Completed | 23
Not completed — Invasive FFR not performed | 21
Not completed — Poor CT Image Quality | 1
Not completed — Invasive FFR Measurement cancelled | 1

BASELINE CHARACTERISTICS:
Groups:
- CCTA: Patients who are scheduled for clinically mandated elective invasive coronary angiography (ICA) at Buffalo General Hospital.
  CCTA Coronary: Diagnostic Test
Arm/Group | CCTA
Number analyzed (Participants) | 52
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 22
  >=65 years | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.7 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 32
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 0
  Unknown or Not Reported | 52
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 17
  Japan | 35
BMI [Mean (Standard Deviation); unit: kg/m^2] | 25.2 (3.9)
Coronary Calcium Score [Mean (Standard Deviation); unit: Coronary Calcium Score] — The Coronary Calcium Score also referred as Agatston score is calculated using a non-contrast computed tomography (CT) scan to measure for the presence and severity of coronary artery disease through identification of calcification in the coronary arteries. Scores can range from 0 to several thousands. The measure is without units. Score categories are as follows: 0 = no coronary disease; 1-100 = low amount of coronary artery disease; 101-400 = moderately elevated score / moderate coronary artery disease; 401-1000 = severely elevated score; >1000 very severely elevated score
  Coronary Calcium Score | 385 (388)
FFR [Count of Participants; unit: Participants]
  FFR>0.8 | 29
  FFR<=0.8 | 23
Diabetes Mellitus [Count of Participants; unit: Participants]
  Yes | 22
  No | 30
Hypertension [Count of Participants; unit: Participants]
  Yes | 33
  No | 19
Hyperlipidemia [Count of Participants; unit: Participants]
  Yes | 38
  No | 14
Smoking [Count of Participants; unit: Participants]
  Former | 16
  Current | 10
  Never | 26
Prior Myocardial Infarction [Count of Participants; unit: Participants]
  Yes | 4
  No | 48
Creatinine [Mean (Standard Deviation); unit: mg/ dl] | 0.83 (0.45)

OUTCOME MEASURES:

1. Primary Outcome: Comparison of CT Based FFR With Invasive FFR, ROC Analysis
Description: Patient CCTA images were imported into Vitrea segmentation software (Vital Images, Minnetonka, MN) for use in the research-based CT based FFR algorithm. The software analyzes four data volumes acquired a 70%, 80%, 90% and 99% of the R-R interval and computes the FFR based on the changes in vessel diameter and computational fluid dynamics. Within the algorithm, the aortic root and three main coronary arteries (LAD, LCX, and RCA) were automatically segmented, and then manually adjusted to obtain accurate centerline and contours. The CT based FFR was calculated and the user adjusted the location of the distal pressure measurement to calculate the CT basedFFR at the same location as Invasive-FFR, two lesion lengths below the distal end of the lesion.
  Area under the Receiver Operator Characteristic were measured where an Invasive FFR<=0.8 was considered positive.
Time Frame: 24 hours
Population: From the total number of patients, nine patients had multi-vessel disease and I-FFR was measured in two vessels. In total I-FFR was measured in: 42 LADs, 11 LCXs and 8 RCAs. Invasive -FFR measurement location was from the ostium to two lesion lengths below the distal throat of the lesion .
Measure: Number (95% Confidence Interval); unit: probability of accurate diagnosis
Units Other Than Participants: Coronary Arteries
Arm/Group | CCTA
Number analyzed (Participants) | 52
Number analyzed (Coronary Arteries) | 61
probability of accurate diagnosis | 0.8 [0.7 to 0.87]

2. Primary Outcome: Comparison of CT Based FFR With Invasive FFR, Correlation Analysis
Description: Patient CCTA images were imported into Vitrea segmentation software (Vital Images, Minnetonka, MN) for use in the research-based CT based FFR algorithm. The software analyzes four data volumes acquired a 70%, 80%, 90% and 99% of the R-R interval and computes the FFR based on the changes in vessel diameter and computational fluid dynamics. Within the algorithm, the aortic root and three main coronary arteries (LAD, LCX, and RCA) were automatically segmented, and then manually adjusted to obtain accurate centerline and contours. The CT based FFR was calculated and the user adjusted the location of the distal pressure measurement to calculate the CT basedFFR at the same location as Invasive-FFR, two lesion lengths below the distal end of the lesion.
  Pearson Correlation between Invasive FFR and CT based FFR was measured
Time Frame: 24 hours
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: correlation coefficient
Units Other Than Participants: Coronary Arteries
Arm/Group | CCTA
Number analyzed (Participants) | 75
Number analyzed (Coronary Arteries) | 61
correlation coefficient | 0.75 [0.62 to 0.85]

3. Primary Outcome: Comparison of CT Based FFR With Invasive FFR, Sensitivity
Description: Patient CCTA images were imported into Vitrea segmentation software (Vital Images, Minnetonka, MN) for use in the research-based CT based FFR algorithm. The software analyzes four data volumes acquired a 70%, 80%, 90% and 99% of the R-R interval and computes the FFR based on the changes in vessel diameter and computational fluid dynamics. Within the algorithm, the aortic root and three main coronary arteries (LAD, LCX, and RCA) were automatically segmented, and then manually adjusted to obtain accurate centerline and contours. The CT based FFR was calculated and the user adjusted the location of the distal pressure measurement to calculate the CT basedFFR at the same location as Invasive-FFR, two lesion lengths below the distal end of the lesion.
  Sensitivity were measured where an Invasive FFR<=0.8 was considered positive. Sensitivity reflects the percentage of true positive cases identified by CT-FFR compared to I-FFR
Time Frame: 24 hours
Population: as for outcome 1
Measure: Number; unit: percentage of true positive cases
Units Other Than Participants: Coronary Arteries
Groups:
- CCTA: Patients who are scheduled for clinically mandated elective invasive coronary angiography (ICA) at Buffalo General Hospital.
  CCTA : Diagnostic Test
Arm/Group | CCTA
Number analyzed (Participants) | 52
Number analyzed (Coronary Arteries) | 61
percentage of true positive cases | 82.61

4. Primary Outcome: Comparison of CT Based FFR With Invasive FFR, Specificity
Description: Patient CCTA images were imported into Vitrea segmentation software (Vital Images, Minnetonka, MN) for use in the research-based CT based FFR algorithm. The software analyzes four data volumes acquired a 70%, 80%, 90% and 99% of the R-R interval and computes the FFR based on the changes in vessel diameter and computational fluid dynamics. Within the algorithm, the aortic root and three main coronary arteries (LAD, LCX, and RCA) were automatically segmented, and then manually adjusted to obtain accurate centerline and contours. The CT based FFR was calculated and the user adjusted the location of the distal pressure measurement to calculate the CT basedFFR at the same location as Invasive-FFR, two lesion lengths below the distal end of the lesion.
  Specificity was measured, where an Invasive FFR<=0.8 was considered positive. Specificity reflects the percentage of true negative cases identified by CT-FFR compared to I-FFR
Time Frame: 24 hours
Population: as for outcome 1
Measure: Number; unit: percentage of of true negative cases
Units Other Than Participants: Coronary Arteries
Arm/Group | CCTA
Number analyzed (Participants) | 52
Number analyzed (Coronary Arteries) | 61
percentage of of true negative cases | 76.32

5. Secondary Outcome: Comparison of CT Based FFR With Bench-top FFR Using 3D Printed Patient Specific Phantoms
Description: CT images were used to measure CT-FFR and to generate patient-specific 3D printed models of the aortic root and three main coronary arteries. Each patient-specific 3D printed model was connected to a programmable pulsatile pump and bench-top FFR (B-FFR) was derived from pressures measured proximal and distal to coronary stenosis using pressure transducers. B-FFR was measured for hyperemic", 500 mL/min by adjusting the model's distal coronary resistance. Linear regression and Pearson correlation was calculated.
Time Frame: 4 weeks from baseline
Population: From the total number of patients, nine patients had multi-vessel disease and Invasive-FFR was measured in two vessels. In total I-FFR was measured in: 42 LADs, 11 LCXs and 8 RCAs. Bench-top FFR was measured at the same locations as Invasive -FFR, from the ostium to two lesion lengths below the distal throat of the lesion .
Measure: Number (95% Confidence Interval); unit: correlation coefficient
Units Other Than Participants: Coronary Arteries
Arm/Group | CCTA
Number analyzed (Participants) | 52
Number analyzed (Coronary Arteries) | 61
correlation coefficient | 0.64 [0.46 to 0.76]

6. Secondary Outcome: Comparison of Bench-top FFR Using 3D Printed Patient Specific Phantoms With Invasive FFR, ROC Analysis
Description: CT images were used to create patient specific 3d-printed phantom. Each patient-specific 3D printed model was connected to a programmable pulsatile pump and benchtop FFR (B-FFR) was derived from pressures measured proximal and distal to coronary stenosis using pressure transducers. B-FFR was measured for hyperemic", 500 mL/min by adjusting the model's distal coronary resistance. Benchtop-FFR was compared with Invasive-FFR. Area under the Receiver Operator Characteristic were measured where an Invasive FFR<=0.8 was considered positive.
Time Frame: 4 weeks from baseline
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: probability of accurate diagnosis
Units Other Than Participants: Coronary Arteries
Arm/Group | CCTA
Number analyzed (Participants) | 52
Number analyzed (Coronary Arteries) | 61
probability of accurate diagnosis | 0.81 [0.64 to 0.91]

7. Secondary Outcome: Comparison of Bench-top FFR Using 3D Printed Patient Specific Phantoms With Invasive FFR, Pearson Correlation
Description: CT images were used to create patient specific 3d-printed phantom. Each patient-specific 3D printed model was connected to a programmable pulsatile pump and benchtop FFR (B-FFR) was derived from pressures measured proximal and distal to coronary stenosis using pressure transducers. B-FFR was measured for hyperemic", 500 mL/min by adjusting the model's distal coronary resistance. Benchtop-FFR was compared with Invasive-FFR. Pearson Correlation factor was calculated.
Time Frame: 4 weeks from baseline
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: correlation coefficient
Units Other Than Participants: Coronary Arteries
Arm/Group | CCTA
Number analyzed (Participants) | 52
Number analyzed (Coronary Arteries) | 61
correlation coefficient | 0.71 [0.56 to 0.81]

8. Secondary Outcome: Comparison of Bench-top FFR Using 3D Printed Patient Specific Phantoms With Invasive FFR, Sensitivity
Description: CT images were used to create patient specific 3d-printed phantom. Each patient-specific 3D printed model was connected to a programmable pulsatile pump and benchtop FFR (B-FFR) was derived from pressures measured proximal and distal to coronary stenosis using pressure transducers. B-FFR was measured for hyperemic", 500 mL/min by adjusting the model's distal coronary resistance. Benchtop-FFR was compared with Invasive-FFR. Sensitivity was measure, where an Invasive FFR<=0.8 was considered positive.Sensitivity reflects the percentage of true positive cases identified by B-FFR compared to I-FFR
Time Frame: 4 weeks from baseline
Population: as for outcome 5
Measure: Number; unit: percentage of true positive cases
Units Other Than Participants: Coronary Arteries
Arm/Group | CCTA
Number analyzed (Participants) | 52
Number analyzed (Coronary Arteries) | 61
percentage of true positive cases | 86.96

9. Secondary Outcome: Comparison of Bench-top FFR Using 3D Printed Patient Specific Phantoms With Invasive FFR, Specificity
Description: CT images were used to create patient specific 3d-printed phantom. Each patient-specific 3D printed model was connected to a programmable pulsatile pump and benchtop FFR (B-FFR) was derived from pressures measured proximal and distal to coronary stenosis using pressure transducers. B-FFR was measured for hyperemic", 500 mL/min by adjusting the model's distal coronary resistance. Benchtop-FFR was compared with Invasive-FFR. Specificity was calculated, where an Invasive FFR<=0.8 was considered positive. Specificity reflects the percentage of true negative cases identified by B-FFR compared to I-FFR
Time Frame: 4 weeks from baseline
Population: as for outcome 5
Measure: Number; unit: percentage of true negative cases
Units Other Than Participants: Coronary Arteries
Arm/Group | CCTA
Number analyzed (Participants) | 52
Number analyzed (Coronary Arteries) | 61
percentage of true negative cases | 97.37

ADVERSE EVENTS:
Time Frame: The participant was observed for 24 hours post CCTA acquisition.
Description: No risk of serious adverse events, mortality, or other adverse events during CCTA scan.
Groups:
- CCTA Coronary: Patients who are scheduled for clinically mandated elective invasive coronary angiography (ICA) at Buffalo General Hospital and Juntendo University, Japan.
  CCTA Coronary: Diagnostic Test
Arm/Group | CCTA Coronary
All-Cause Mortality (participants affected / at risk) | 0/52
Serious Adverse Events (participants affected / at risk) | 0/52
Other Adverse Events (participants affected / at risk) | 0/52

LIMITATIONS AND CAVEATS:
Operators were not blinded to the invasive-FFR results at the time of calculating the CT based FFR and Bench-top measurements

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Informed Consent Form (2019-01-15): https://cdn.clinicaltrials.gov/large-docs/42/NCT03149042/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2019-09-24): https://cdn.clinicaltrials.gov/large-docs/42/NCT03149042/Prot_SAP_001.pdf